CLINICAL TRIAL: NCT06339099
Title: Enhancing Gross Motor Function and Knee Extensor Strength During Loaded Gait Training in Children with Bilateral Spastic Cerebral Palsy: a Randomized Controlled Trial
Brief Title: Loaded Gait Training on Gross Motor Function in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amina Awad,PhD, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002489
Record Dates: First submitted 2024-03-18; First posted 2024-04-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy
Keywords: Bilateral spastic CP,; Gross motor function; Knee extensor strength; Loaded gait training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Children were randomly assigned into two equal groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinding. Parents were also blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control arm (Experimental): The control group (n=26) received a conventional physical therapy program.
  Interventions: Other: Conventional physical therapy program
- Intervention arm (Active Comparator): The intervention group (n=26) received conventional physical therapy program and loaded gait training.
  Interventions: Other: Conventional physical therapy program; Other: Loaded gait training

INTERVENTIONS:
Other: Conventional physical therapy program — This program included active resisted strengthening exercises for pelvis girdle and lower limb muscles, stretching exercises of tight muscles of lower limbs; hip flexors, hamstrings and calf muscle, balance activities from standing and walking and gait training exercises.
Other: Loaded gait training — An extra weight was added around the distal legs during gait training in the intervention group. This weight began at 0.5 kg and was gradually increased every two weeks to a maximum of 2 kg
  Arms: Intervention arm

SUMMARY:
A randomized controlled trial aimed to evaluate the additional effect loaded gait training to conventional physical therapy program on gross motor function and the knee extensors strength in children with bilateral spastic cerebral palsy. Children were divided randomly into two equal groups. The control group received a conventional physical therapy program, while the intervention group received the same program plus loaded gait training. Gross motor functions and knee extensor strength were measured.

DETAILED DESCRIPTION:
A randomized controlled trial aimed to evaluate the additional effect loaded gait training to conventional physical therapy program on gross motor function and the knee extensors strength in children with bilateral spastic cerebral palsy (CP).

52 children with bilateral spastic CP, aged 5 to 7 years, were divided randomly into two equal groups. The control group received a conventional physical therapy program, while the intervention group received the same program plus loaded gait training 3 times per week for an hour for 3 months.

Gross motor functions were measured by the Gross Motor Function Measure Scale-88 (GMFM-88); standing and walking domains, while knee extensor strength was measured by a hand-held dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Age: five to seven years old, classified as levels II and III on the GMFCS.
* Spasticity grade from 1+ to 2 based on the Modified Ashworth scale.
* Able to understand and follow verbal commands and instructions (with a score above 80 on the Stanford Binet Intelligence Scale).

Exclusion Criteria:

* Genetic or metabolic disorders.
* Brain tumours.
* Musculoskeletal dysfunction that would interfere with our intervention (e.g. tightness of the posterior knee joint capsule that causes passive knee extension lag, or fixed contracture of the knee joint).
* Surgical intervention in the lower limbs within the preceding 12 months.
* Botulinum toxin injections in lower limb muscles within the last six months.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Gross motor function | 1 year
  Gross Motor Function Measure Scale-88 (GMFM-88); standing and walking domains.
knee extensor strength | 1 year
  Knee extensor strength was measured by a hand-held dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Radwa S Abdul-Rahman, PhD, Principal Investigator — Faculty of Physical Therapy, Cairo University, Egypt
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No